CLINICAL TRIAL: NCT06586905
Title: A Cross-sectional Investigational Study to Evaluate the Sensitivity, Specificity, and Utility of the MedMira Inc. Multiplo® Complete Syphilis (TP/nTP) Antibody Test (POCT) to Diagnose Infectious Syphilis in Participants Attending the Sexual Health Clinic in Ottawa, Ontario. The MedMira Inc. Multiplo® Complete Syphilis (TP/nTP) Antibody Test is Authorized for Investigational Use.
Brief Title: A Cross-sectional Investigational Study to Evaluate the Sensitivity, Specificity, and Utility of the MedMira Inc. Multiplo® Complete Syphilis (TP/nTP) Antibody Test (POCT) to Diagnose Infectious Syphilis in Participants Attending the Sexual Health Clinic in Ottawa, Ontario.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MedMira Laboratories Inc. (Industry)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REB 2023-034P
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Syphilis; Treponema Pallidum
Keywords: Syphilis; TP/nTP; Multiplo Complete Syphilis (TP/nTP) Antibody Test; MedMira; Treponema pallidum; rapid test; point of care
MeSH Terms: conditions — Syphilis; Treponemal Infections | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiplo Complete Syphilis (TP/nTP) Antibody Test (Experimental): Participants are tested with investigational devices and conventional syphilis serology tests
  Interventions: Device: Medical Device

INTERVENTIONS:
Device: Medical Device — Multiplo Complete Syphilis (TP/nTP) Antibody Test

SUMMARY:
Due to the recent resurgence of infectious syphilis in Canada and the changing epidemiology of the disease to involve heterosexuals and females of child bearing age leading to a record number of congenital syphilis cases and stillbirths, the demand of a rapid test such as POCT that can be used at the place and time that front-line public health workers meet the at risk population is getting louder. Indeed during a number of federal, provincial and territorial meetings on the control of syphilis outbreaks in Canada, requests for POCT to detect syphilis infections have repeatedly come up. However, before a POCT can be widely used, research to find out if it is accurate and reliable is necessary. This study is designed to test the performance of the MedMira Inc. Multiplo® Complete Syphilis (TP/nTP) Antibody Test (POCT) (MedMira Inc., Halifax, Nova Scotia) in an urban clinic (Sexual Health Clinic) in Ottawa, Ontario, Canada and compare its performance in parallel with the usual testing method (the gold standard, i.e. conventional syphilis serology testing).

ELIGIBILITY:
Inclusion Criteria:

* Individuals attending the Clinic for routine sexual health care and requiring syphilis testing as part of this care, who are able to provide informed consent and are a minimum 16 years of age are eligible for this study. This includes patients attending the Clinic for follow-up appointments following diagnosis with syphilis infection. Those who have had other STIs in the past, or being suspected of having other STIs, are not excluded as long as testing for syphilis is part of the care provided to them. Once it has been determined that the exclusion criteria does not apply to a patient, the recruitment of participants will be offered without other pre-selection criteria unless there may be other unforeseeable circumstances arising, such as shortage of Clinic staff or large numbers of patients in attendance.

Exclusion Criteria:

* Those who, at the discretion of the HCPs/research co-ordinator, appear intoxicated and/or with extreme distress, or confused, will be excluded from this research because they would not be able to provide informed consent to participate, as well as those below the age of 16 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
To determine the accuracy of Multiplo Complete Syphilis (TP/nTP) Antibody Test | 1 patient visit of appoximately 30 minutes
  For each enrolled subject, Multiplo Complete Syphilis (TP/nTP) Antibody Test will be used to test fingerstick whole blood from the patient. A venipuncture whole blood sample will also be drawn from the patient and will be tested using conventional serological testing methods to determine patient status.

CONTACTS AND LOCATIONS:
Locations (1):
- Sexual Health Clinic, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Byrne P, Dillabough R, Whyte K, Orser L, Tran V, Duvvuri VR, Tsang R. Evaluating the MedMira Multiplo(R) Complete Syphilis (TP/nTP) antibody test in a sexually transmitted infection clinic in Ottawa, Canada: increased rapid diagnosis and improved antibiotic stewardship. BMC Infect Dis. 2025 Dec 8;26(1):48. doi: 10.1186/s12879-025-12263-w. PMID 41361278